CLINICAL TRIAL: NCT05310955
Title: Discussion on the Intervention Effect of Shen-based Qigong Exercise on Residual Symptoms of Schizophrenia Based on the Theory of "Heart Dominating Mind" and "Body-spirit Syncretism" in Traditional Chinese Medicine
Brief Title: Intervention Effect of Shen-based Qigong Exercise on Residual Symptoms of Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YSF2021-59
Record Dates: First submitted 2022-02-22; First posted 2022-04-05 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): daily rehabilitation interventions
  Interventions: Other: daily rehabilitation interventions
- Interventional group (Experimental): daily rehabilitation interventions and shen-based Qigong exercise
  Interventions: Other: daily rehabilitation interventions; Other: shen-based Qigong exercise

INTERVENTIONS:
Other: daily rehabilitation interventions — including Naikan therapy, Morita therapy, group art therapy, group painting therapy
Other: shen-based Qigong exercise — a 12-week intervention of shen-based Qigong exercise : exercise 5 days a week, about 30 minutes a day
  Arms: Interventional group

SUMMARY:
The purpose of this study is to observe the intervention effect of shen-based Qigong exercise on residual symptoms of schizophrenia.

DETAILED DESCRIPTION:
Shen-based Qigong exercise is a new kind of health-care Qigong exercise based on the theory of traditional Chinese medicine, aiming at the characteristics of schizophrenia. In this study, a randomized controlled trial was conducted to observe the rehabilitation effect of this new exercise on residual symptoms of schizophrenic patients. Questionnaire, test and other experimental materials were used to evaluate the intervention effect of 12-week shen-based Qigong exercise on psychiatric symptoms, cognitive function, quality of life and social function of schizophrenic patients. At the same time, the related physical function and cardiac function indexes were used to evaluate the physical and cardiac rehabilitation effects of the exercise on patients from the aspects of "body" and "heart", so as to verify whether Qigong exercise has the effects of adjusting body and heart.

ELIGIBILITY:
Inclusion Criteria:

1. Han Chinese population
2. age ≥ 18 years
3. education level ≥ 6 years, can fill in the questionnaire independently, have enough audio-visual level to complete the necessary examination
4. assessed by MINI 7.0 and satisfied with the diagnostic criteria for schizophrenia based on the Diagnostic and Statistical Manual of Mental Disorders, fifth edition(DSM-5)
5. patients with schizophrenia residing in the rehabilitation ward, without relapse in the past 6 months
6. residual negative symptoms, with at least one item ≥ 2 on the negative subscale of PANSS (N1-N7)
7. taking second generation antipsychotics
8. no training history of traditional Chinese exercises
9. agreement to participate in the study and willing to give written informed consent

Exclusion Criteria:

1. having severe physical diseases such as cardiovascular, lung, liver, kidney, and hematopoietic diseases
2. satisfied with the diagnostic criteria for other mental disorders based on DSM-5
3. having alcohol or substance abuse/dependence
4. having mental retardation(WAIS<70) and/or severe cognitive impairment(MMSE<24)
5. having visual and / or hearing problems, unable to complete the relevant test
6. electroconvulsive or repetitive transcranial magnetic stimulation(rTMS) therapy in the past 3 months
7. currently enrolled or participated in other clinical studies in the past 3 months
8. participating in regular exercise training in the past 6 months
9. failure to sign or refuse to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
change of the Scale for the Assessment of Negative Symptoms (SANS) | Change from Baseline at 3 months
  Negative symptoms will be evaluated using the Scale for the Assessment of Negative Symptoms (SANS). The scale made up for the lack of attention to negative symptoms in previous psychiatric rating scales. It contains five subscales: affective blunting, alogia, avolition/apathy, anhedonia/asociality, and attention. A total of 24 items were scored at 6 levels for each item.

SECONDARY OUTCOMES:
change of Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Change from Baseline at 3 months
  RBANS will be used to assess global cognitive function. RBANS yields scaled scores for 5 cognitive domains and shows a good effect in cognitive assessment of patients with schizophrenia.
change of event-related potential P300 (ERP P300) | Change from Baseline at 3 months
  ERP P300 will be used to assess global cognitive function. ERP P300 is an endogenous cognitive component related to high-level psychological activities such as attention, memory, feeling, learning and reasoning. It has good stability and can reflect the level of cognitive function from different aspects.

OTHER OUTCOMES:
change of n-back task | Change from Baseline at 3 months
  Specific cognitive domain--working memory will be assessed by n-back task. N-back task paradigm is the most classical paradigm in working memory research.
change of 36-item Short Form Health Survey（SF-36） | Change from Baseline at 3 months
  36-item Short Form Health Survey（SF-36）will be used to assess the health-related quality of life of patients. SF-36 is one of the most commonly used standardized measurement tools for quality of life in the world, including eight subscales, a total of 36 items, involving physical and mental health.
change of Social-Adaptive Functioning Evaluation (SAFE) | Change from Baseline at 3 months
  Social functions will be assessed using Social-Adaptive Functioning Evaluation (SAFE). SAFE can evaluate the social adaptation function of patients with mental disorders over 18 years old. It has a total of 19 items, divided into basic life skills, advanced life skills, social skills and communication skills in four areas; each item 0-4 score, the higher the score, the more serious the damage.
change of the Scale for the Assessment of Positive Symptoms (SAPS) | Change from Baseline at 3 months
  Positive symptoms will be evaluated using the Scale for the Assessment of Positive Symptoms (SAPS). SAPS measures positive symptoms on a 34 item, 6-point scale, a total of 170 points. Items are listed under hallucinations, delusions, bizarre behavior, and positive formal thought disorder.
change of heart rate variability (HRV) | Change from Baseline at 3 months
  Heart rate variability (HRV) will be used as the evaluation index for cardiac function. HRV is a widely used non-invasive tool for evaluating cardiac autonomic nerve function.
change of height | Change from Baseline at 3 months
  Height will be measured using a height ruler, expressed in meters.
change of weight | Change from Baseline at 3 months
  Weight will be measured using a weighting scale, expressed in kilograms.
change of waistline | Change from Baseline at 3 months
  Waistline will be measured using a flexible rule, expressed in centimeters.
change of blood pressure | Change from Baseline at 3 months
  Blood pressure will be measured using a sphygmomanometer, expressed in millimeter of mercury.
change of gait data | Change from Baseline at 3 months
  Acquire gait data in a quiet, well-lit room. Specify the walking area to guide the participants to complete the walking cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Fan, Study Chair — Shanghai Mental Health Center; Xiaodan Liu, Study Chair — School of Rehabilitation Science, Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Shen H, Lian A, Wu Y, Zhou J, Liu Y, Zhu L, Zhang Y, Yi Z, Liu X, Fan Q. Shen-based Qigong Exercise improves cognitive impairment in stable schizophrenia patients in rehabilitation wards: a randomized controlled study. BMC Psychiatry. 2024 Nov 13;24(1):796. doi: 10.1186/s12888-024-06146-8. PMID 39538216
- [Derived] Lian A, Fan Q, Wang W, Liu Q, Shi J, Zhuang M, Li Y, Liu X. Effect of 12-week shen-based qigong exercise on the residual symptoms of schizophrenia: Study protocol for a single-centre randomised controlled trial. Contemp Clin Trials Commun. 2023 Oct 3;36:101214. doi: 10.1016/j.conctc.2023.101214. eCollection 2023 Dec. PMID 37842323